CLINICAL TRIAL: NCT03314363
Title: MEtabolic Consequences of Continuous Renal Replacement Therapy and Impact on Indirect cAlorimetry Study
Brief Title: Plasma CO2 Removal Due to CRRT and Its Influence on Indirect Calorimetry
Acronym: MECCIAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Elisabeth De Waele, Principal Investigator, clinical professor, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B.U.N. 143201731636
Record Dates: First submitted 2017-07-03; First posted 2017-10-19 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Continuous Renal Replacement Therapy; CO2 Removal; Nutrition Poor; Acute Renal Failure
Keywords: Calorimetry, Indirect; respiratory dialysis
MeSH Terms: conditions — Malnutrition; Acute Kidney Injury | interventions — Trace Elements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- all patients (Other): Classic CRRT with citrate predilution
  Interventions: Diagnostic Test: blood gas analysis under citrate predilution; Device: filter replacement; Device: IC; Drug: NaCl predilution; Diagnostic Test: blood gas analysis under NaCl predilution; Drug: double ultrafiltration; Diagnostic Test: blood gas analysis under citrate predilution and double ultrafiltration rate; Dietary Supplement: pause and restart nutritional therapy; Diagnostic Test: evolution of vitamin and trace elements

INTERVENTIONS:
Diagnostic Test: blood gas analysis under citrate predilution — blood gas analysis of blood on different sample points and dialysis fluid
Device: filter replacement — Using local protocol: stop and disconnect CRRT, replace filter and reconnect and restart CRRT.
Device: IC — monitor patients during the whole study period with indirect calorimetry
Drug: NaCl predilution — Replace citrate predilution with NaCl
Diagnostic Test: blood gas analysis under NaCl predilution — repeat blood gas analysis of blood on different sample points and dialysis fluid
Drug: double ultrafiltration — double the ultrafiltration fluid by augmenting post dilution fluid and keeping ultrafiltration at the same rate.
Diagnostic Test: blood gas analysis under citrate predilution and double ultrafiltration rate — repeat blood gas analysis of blood on different sample points and dialysis fluid
Dietary Supplement: pause and restart nutritional therapy — pause parenteral and enteral nutrition before indirect calorimetry is performed. and restart after first blood analysis for vitamine status
Diagnostic Test: evolution of vitamin and trace elements — blood analysis for vitamin and trace elements. Perform this blood analysis after restart of CRRT but before restart of nutritional therapy, 30 minutes after restart of nutritional therapy and 24h after restart of nutritional therapy.

SUMMARY:
The aim of the present study is to assess the metabolic impact of Continuous Renal Replacement Therapy and overview the obstacles and important factors compromising the use of Indirect Calorimetry in CRRT and suggest a model to overcome these issues.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) complicates a critical illness from 13% up to 78%, needing renal replacement therapy (RRT) up to10 % of all patients in the intensive care unit (ICU). Both intermittent (IRRT) and continuous renal replacement therapy (CRRT) are used. The advantage of the latter is that it has lesser influence on hemodynamics and is better tolerated in critical ill patients.

Another complication during their stay is the inability to feed themselves. Nutrition is a cornerstone in the care for the critical ill and should be started within 3 days of admission to the intensive care unit. To optimize a nutritional prescription, protein and energy targets need to be defined. Predicting formulae based on anthropometric measures and other parameters can be used to calculate the caloric need but indirect calorimetry (IC) remains the gold standard. Caloric need can be derived from Energy expenditure which is calculated with the Weir's equation using carbon dioxide (CO2) production (VCO2) and oxygen (O2) consumption (VO2). Therefore, it is underestimated if CO2 is lost through other means than the normal respiratory route. Hence one of the contra-indications of IC is CRRT.

The totalCO2 (tCO2) travels through the vascular structures within the red blood cells or inside plasma. There, most of the content has 3 different forms: as physically dissolved CO2, bicarbonate, and carbamino compounds. These compounds are in equilibrium with each other. During RRT, a potential loss of CO2 and its different forms may occur due to ultrafiltration in the dialysate. No large trials were conducted trying to quantify this loss nor identifying the determining factors which can be used to predict this loss. Indeed, one author even found a gain in tCO2 of the blood during dialysis with acetate. Trisodiumcitrate is used as an anticoagulant during CRRT. It is a weak base and due to pH change may alter the equilibrium of the Henderson-Hasselbalch equation and thus influence the balance between CO2 and HCO3- and its extraction through CRRT.

Although indirect calorimetry in the intensive care unit has been evaluated during CRRT, the loss of tCO2was not considered. The investigators explored the possibility to predict and easily calculate this CO2 exchange so IC can be used during CRRT.

ELIGIBILITY:
Inclusion Criteria:

* AKI requiring CRRT
* Patient on CRRT who's filter you want to change
* Expected stable patient during the test ( +- 2h) evaluated at discretion of physician :

  * No alteration in medication
  * Stable respiratory settings where no change in conditions is expected. If possible, controlled mode ventilation is preferred.
  * Expected stable pH and lactate
  * no intervention will be made on patient (transport/washing/physiotherapy/…)
  * no alterations on settings of CRRT is expected to be made.
* Maximal respiratory settings: max FiO2: 60% / max inspiratory plateau pressure 30 mmHg/max tidal volumes 8ml/kg
* pH between 7,30-7,50, lactate levels <2,0
* starting settings CRRT with citrate:

  * Blood pump flow: 150 ml/min
  * Predilution ( citrate): 1500-2300ml/h
  * Dialysate dose: 25-40 ml/kg/h
  * ultrafiltration: 0-300 ml /h
  * Substitution: NaCl 300-800 ml/h or B22: 400-2000 ml/h

Exclusion Criteria:

* Pregnancy / lactation
* Contra-indications for the use of indirect calorimetry as stated by the AARC (FiO2>60%, chest tubes)
* Severe hemodynamic or ventilator instability.
* CRRT modalities unusual to daily clinical ICU practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
change in CO2 flow and O2 flow on different sample points of CRRT | 2hours
  CO2 flow and O2 flow ( ml/min) will be compared between the different sample points on CRRT with and without citrate.
  CO2 flow and O2 flow is calculated by multiplying fluid flow ( ml/min) on different sample points of CRRT with CO2 content or O2 content of fluid on respective sample points during CRRT with and without Citrate.
REE change due to CRRT | 2hours
  REE ( Kcal) will be measured during the whole procedure using IC. REE will be measured during CRRT. citrate wil be replaced by NaCl 0,9% fluid and REE will be measured. After this, CRRT will be stopped and REE will be measured. The difference in REE during CRRT with and without citrate and without CRRT will be calculated and compared.
  REE is calculated using the weir equation and VO2, VCO2. VO2 and VCO2 is calculated using FiO2, FeO2, FiCO2, FeCO2 and VE.
does change in CO2 flow and O2 flow on different sample points of CRRT correlate with VCO2 and VO2 change due to CRRT with or without citrate | 2 hours
  VCO2 and VO2 change due to CRRT and due to citrate will be correlated with change in CO2 and O2 flow of fluids passing through CRRT with or without citrate.
Are vitamins and trace elements sufficiently supplemented with standard nutritional therapy during CRRT | 24hours
  blood analysis for concentrations of Vitamin A, B1, B6, B9, B12, C, D, E ; trace elements selenium, zinc, copper, chrome; and cholesterol and triglyceride

SECONDARY OUTCOMES:
VCO2 and VO2 change due to CRRT with or without citrate | 2 hours
  VCO2 and VO2 ( ml/min) will be measured during the whole procedure using IC. VCO2 and VO2 will be measured during CRRT with citrate. citrate wil be replaced by NaCl 0,9% fluid and VCO2 and VO2 will be measured. After this, CRRT will be stopped and VCO2 and VO2 will be measured. The difference in VCO2 and VO2 during CRRT with or without citrate and without CRRT will be calculated and compared. VO2 and VCO2 is calculated using FiO2, FeO2, FiCO2, FeCO2 and VE.
FiO2, FeO2, FiCO2 and FeCO2 change due to CRRT with or without citrate | 2hours
  FiO2, FeO2, FiCO2 and FeCO2 ( %) will be measured during the whole procedure using IC. FiO2, FeO2, FiCO2 and FeCO2 will be measured during CRRT with citrate. citrate wil be replace by NaCl0,9% fluid and FiO2, FeO2, FiCO2 and FeCO2 will be measured. After this CRRT will be stopped and FiO2, FeO2, FiCO2 and FeCO2 will be measured. The difference in FiO2, FeO2, FiCO2 and FeCO2 during CRRT with or without citrate and without CRRT will be calculated.
VE change due to CRRT with or without citrate | 2hours
  VE( ml/min) will be measured during the whole procedure using IC. VE will be measured during CRRT with citrate. citrate wil be replace by NaCl0,9% fluid and VE will be measured. After this CRRT will be stopped and VE will be measured. The difference in VE during CRRT with or without citrate and without CRRT will be calculated.
change in CO2 and O2 content of fluid passing through CRRT | 2hours
  using blood gas analyser, CO2 content and O2content ( mmol/L)of fluid on different sample points in extracorporeal circuit of CRRT with or without citrate will be analysed and compared.
change in bicarbonate content of fluid passing through CRRT | 2hours
  using blood gas analyser, bicarbonate ( mmol/L) of fluid on different sample points in extracorporeal circuit of CRRT with or without citrate will be analysed and compared.
change in pH change of fluid passing through CRRT | 2hours
  using blood gas analyser, pH of fluid on different sample points in extracorporeal circuit of CRRT with or without citrate will be analysed and compared
change in pCO2 and pO2 change of fluid passing through CRRT | 2hours
  using blood gas analyser, pCO2 and pO2 (mmHg) of fluid on different sample points in extracorporeal circuit of CRRT with or without citrate will be analysed and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth De Waele, Phd, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- universitair ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Case J, Khan S, Khalid R, Khan A. Epidemiology of acute kidney injury in the intensive care unit. Crit Care Res Pract. 2013;2013:479730. doi: 10.1155/2013/479730. Epub 2013 Mar 21. PMID 23573420
- [Result] Metnitz PG, Krenn CG, Steltzer H, Lang T, Ploder J, Lenz K, Le Gall JR, Druml W. Effect of acute renal failure requiring renal replacement therapy on outcome in critically ill patients. Crit Care Med. 2002 Sep;30(9):2051-8. doi: 10.1097/00003246-200209000-00016. PMID 12352040
- [Result] Rabindranath K, Adams J, Macleod AM, Muirhead N. Intermittent versus continuous renal replacement therapy for acute renal failure in adults. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003773. doi: 10.1002/14651858.CD003773.pub3. PMID 17636735
- [Result] Singer P, Berger MM, Van den Berghe G, Biolo G, Calder P, Forbes A, Griffiths R, Kreyman G, Leverve X, Pichard C, ESPEN. ESPEN Guidelines on Parenteral Nutrition: intensive care. Clin Nutr. 2009 Aug;28(4):387-400. doi: 10.1016/j.clnu.2009.04.024. Epub 2009 Jun 7. PMID 19505748
- [Result] Wichansawakun S, Meddings L, Alberda C, Robbins S, Gramlich L. Energy requirements and the use of predictive equations versus indirect calorimetry in critically ill patients. Appl Physiol Nutr Metab. 2015 Feb;40(2):207-10. doi: 10.1139/apnm-2014-0276. Epub 2014 Oct 27. PMID 25610953
- [Result] Oshima T, Berger MM, De Waele E, Guttormsen AB, Heidegger CP, Hiesmayr M, Singer P, Wernerman J, Pichard C. Indirect calorimetry in nutritional therapy. A position paper by the ICALIC study group. Clin Nutr. 2017 Jun;36(3):651-662. doi: 10.1016/j.clnu.2016.06.010. Epub 2016 Jun 22. PMID 27373497
- [Result] Honore PM, De Waele E, Jacobs R, Mattens S, Rose T, Joannes-Boyau O, De Regt J, Verfaillie L, Van Gorp V, Boer W, Collin V, Spapen HD. Nutritional and metabolic alterations during continuous renal replacement therapy. Blood Purif. 2013;35(4):279-84. doi: 10.1159/000350610. Epub 2013 May 8. PMID 23689499
- [Result] AARC clinical practice guideline. Metabolic measurement using indirect calorimetry during mechanical ventilation. American Association for Respiratory Care. Respir Care. 1994 Dec;39(12):1170-5. No abstract available. PMID 10146137
- [Result] Bosch JP, Glabman S, Moutoussis G, Belledonne M, von Albertini B, Kahn T. Carbon dioxide removal in acetate hemodialysis: effects on acid base balance. Kidney Int. 1984 May;25(5):830-7. doi: 10.1038/ki.1984.97. PMID 6433099
- [Result] Scheinkestel CD, Kar L, Marshall K, Bailey M, Davies A, Nyulasi I, Tuxen DV. Prospective randomized trial to assess caloric and protein needs of critically Ill, anuric, ventilated patients requiring continuous renal replacement therapy. Nutrition. 2003 Nov-Dec;19(11-12):909-16. doi: 10.1016/s0899-9007(03)00175-8. PMID 14624937
- [Result] Wu C, Wang X, Yu W, Li P, Liu S, Li J, Li N. Short-term consequences of continuous renal replacement therapy on body composition and metabolic status in sepsis. Asia Pac J Clin Nutr. 2016;25(2):300-7. doi: 10.6133/apjcn.2016.25.2.29. PMID 27222413
- [Derived] Jonckheer J, Spapen H, Debain A, Demol J, Diltoer M, Costa O, Lanckmans K, Oshima T, Honore PM, Malbrain M, De Waele E. CO2 and O2 removal during continuous veno-venous hemofiltration: a pilot study. BMC Nephrol. 2019 Jun 17;20(1):222. doi: 10.1186/s12882-019-1378-y. PMID 31208356